CLINICAL TRIAL: NCT02634385
Title: Zero Ischemia Laparoscopic Partial Nephrectomy in Combination With Superselective Renal Artery Embolization for Small Renal Masses: A Feasibility Trial
Brief Title: Zero Ischemia Laparoscopic Partial Nephrectomy
Acronym: ZILPAREMZ
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: No funding to start project.
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Anil Kapoor, MD, FRCSC, McMaster University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZILPAREMBZ14
Record Dates: First submitted 2014-10-10; First posted 2015-12-18 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Small Renal Mass

ARMS (1):
- Small Renal Mass (No Intervention): Patient's with a small renal mass will be undergoing embolization prior to laparoscopic partial nephrectomy.
  Interventions: Procedure: Renal Artery Embolization; Procedure: Partial Nephrectomy (Surgical Resection)

INTERVENTIONS:
Procedure: Renal Artery Embolization — Patients will be receiving embolization prior to planned partial nephrectomy.
Procedure: Partial Nephrectomy (Surgical Resection) — Patients will be undergoing planned partial nephrectomy post embolization.

SUMMARY:
Laparoscopic partial nephrectomy (LPN) is often reserved for patients with a small peripheral tumour, in the hands of an experienced surgeon since it demands a high degree of endoscopic skill. Renal vessel clamp for vascular control is a required step during standard LPN. However, this creates a time limiting step for the surgeon and induces renal injury via warm ischemia and reperfusion injury. This novel approach can substantially reduce renal injury during LPN via superselective embolization of level II renal arteries pre-operatively. This technique facilitates the performance of a clamp-less, zero-ischemia LPN, significantly simplifying the procedure by remove time thresholds within which to perform tumor excision. The preliminary results are promising; however, there is a need for further corroboration of their results, in addition to a randomized controlled trial comparing this modified, zero ischemia technique with standard LPN.

DETAILED DESCRIPTION:
The potential utility of a zero ischemia, laparoscopic, partial nephrectomy portends significant implications for both the surgeon and patient. Firstly, the technical difficulty of a partial nephrectomy will be reduced to a more achievable level owing mainly to the removal of a time limit on surgical resection. With the blood flow halted to downstream tissue containing the renal neoplasm from preoperative embolization, resection can be made to the tumor without clamping of the main renal arteries. This minimizes the ischemic time to non-neoplastic renal tissue, allowing for a renal protective effect. Without the need for clamping, the overall surgical operative time is drastically reduced. With excision made at the ischemic tissue, intra-operative bleeding and ease can be achieved. More surgeons can ultimately attempt at LPN by removing the single most limiting surgical factor, warm ischemic time.

ELIGIBILITY:
Inclusion Criteria:

* T1a renal cell carcinomas diagnosed by ultrasonography (US), computed tomography (CT) or fine needle aspiration
* tumor size <4cm in diameter
* predominant exophytic growth
* intraparenchymal depth no greater than 1.5cm, with a minimum distance of 5mm from the urinary collecting system

Exclusion Criteria:

* predominant endophytic nature (depth </= 1.5 cm)
* nearness (<0.5cm) of the tumor to the urinary collecting system
* multiple ipsilateral lesions
* pregnancy
* allergy to intravenous contrast dye
* absolute contraindications to surgical intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11; Primary Completion 2016-04 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Extirpative time | Duration of Surgical Procedure
  From initial renal tissue breach until completion of bolster placement. Calculated in minutes.
Warm ischemia time | Duration of Surgical Procedure
  From renal vessel clamping to unclamping during nephrectomy (only if clamping has occurred). Calculated in minutes.
Mean estimated blood loss (measured in ml) | Duration of Surgical Procedure
  From the start of procedure (Nephrectomy), until the end of the procedure.

SECONDARY OUTCOMES:
Mean hospital stay | 2-10 Days
  Date admitted for procedure until date of discharge. Measure in calendar days.
Blood transfusions | From date of pre-op up to 6 months post-op
  Prior to Embolization procedure and pre and post-nephrectomy.
Conversion to other type of surgery (i.e. Radical Nephrectomy) | Duration of Surgical Procedure
  Minutes from the start of procedure (Nephrectomy).
Identification of other complications (i.e. readmission, arteriovenous malformations) | Up to 24 months post-operatively.
  Complications will be monitored after patient is discharged up until two years post-operatively.
Overall survival rates | Up to 24 months post-operatively.
  Follow-up will be monitored.
Pathological Results (% of negative margins and benign versus malignant tumours). | 7 to 14 days post nephrectomy.
  Pathology results are usually not released until 7-14 days post nephrectomy.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Healthcare Hamilton - McMaster Institute of Urology, Hamilton, Ontario, Canada